CLINICAL TRIAL: NCT03462329
Title: Impact of Patient's Pretreatment Expectations on Treatment Outcome of Early Lyme Borreliosis
Brief Title: Patient's Pretreatment Expectations About Post-Lyme Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, MD, PhD, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pretreatment expectations
Record Dates: First submitted 2018-02-19; First posted 2018-03-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Erythema Migrans
Keywords: Post-Lyme symptoms; Pretreatment expectations
MeSH Terms: conditions — Glossitis, Benign Migratory | interventions — Anti-Bacterial Agents; BID protein, human

STUDY DESIGN:
Intervention Model Description: Patients will evaluate their pre-treatment expectations about treatment outcome of erythema migrans.
  Nonspecific symptoms will be assessed in patients and control subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with erythema migrans (Active Comparator): Patients will be treated with antibiotics for Lyme disease.
  Interventions: Drug: Antibiotics (preferentially oral doxycycline 100 mg bid)
- controls (No Intervention): Control subjects will not be given antibiotics.

INTERVENTIONS:
Drug: Antibiotics (preferentially oral doxycycline 100 mg bid) — Patients will be treated with antibiotics for Lyme disease.
  Arms: patients with erythema migrans

SUMMARY:
The investigators will focus on pretreatment expectations of patients with early Lyme disease manifested as erythema migrans with the aim of assessing the association between pretreatment expectations quantified with a questionnaire and treatment outcome quantified with the presence of post-Lyme symptoms. Furthermore, the investigators will compare the prevalence of nonspecific symptoms among patients and among age-matched controls without a history of Lyme borreliosis.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans

Exclusion Criteria:

* pregnancy or lactation
* immunocompromised
* taking antibiotic with antiborrelial activity within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 14 days postenrollment in patients treated for erythema migrans | Study point: at 14 days post-enrollment.
  At follow-up at 14 days patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 2 months postenrollment in patients treated for erythema migrans | Study point: at 2 months post-enrollment.
  At follow-up at 2 months patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 6 months postenrollment in patients treated for erythema migrans | Study point: at 6 months post-enrollment.
  At follow-up at 6 months patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 12 months postenrollment in patients treated for erythema migrans | Study point: at 12 months post-enrollment.
  At 12 months patients will be examined physically and will be asked an open question about health-related symptoms.
  Symptoms that will newly develop or worsen since the onset of erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms. Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.

SECONDARY OUTCOMES:
Change in occurrence of nonspecific symptoms from baseline to 6 months and to 12 months post-enrollment in patients with erythema migrans and control subjects | Study points will be: at enrollment, at 6, and at 12 months post-enrollment.
  Patients will complete a written questionnaire asking whether they had had any of 8 nonspecific symptoms (fatigue, arthralgias, headache, myalgias, paresthesias, memory difficulties, concentration difficulties, irritability) within the preceding week. Control subjects will complete the same 8-symptom questionnaire as the patients within 14 days of the examination date of the corresponding patient at enrollment, and again at 6 and 12 months. Patients and controls will grade the severity of each individual symptom on a 10-cm visual analogue scale (10 = most severe).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical center Ljubljana, Ljubljana, Slovenia